CLINICAL TRIAL: NCT04988152
Title: A Phase I, Single-blind, Randomized, Single-dose Clinical Pharmacology Study to Investigate the Pharmacokinetics, Safety, and Tolerability of Sotrovimab vs Placebo by Intravenous or Intramuscular Administration in Healthy Japanese and Caucasian Participants
Brief Title: A Study to Investigate the PK, Safety, and Tolerability of Sotrovimab vs Placebo Administered IV or IM in Japanese and Caucasian Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vir Biotechnology, Inc. (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: VIR-7831-5009; GSK Study 217653 (Other: GlaxoSmithKline)
Record Dates: First submitted 2021-07-26; First posted 2021-08-03 (Actual); Results first posted 2024-06-07 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2022-09

CONDITIONS: Covid19
Keywords: SARS-CoV-2 coronavirus; coronavirus disease 2019; COVID-19; Japanese pharmacokinetics
MeSH Terms: conditions — COVID-19 | interventions — sotrovimab

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1 Sotrovimab intravenous infusion, single dose (Experimental)
  Interventions: Biological: sotrovimab
- Part 1 Volume-matched placebo, intravenous infusion (Placebo Comparator)
  Interventions: Other: Placebo to Biologic
- Part 2 Sotrovimab intramuscular injection, single dose (Experimental)
  Interventions: Biological: sotrovimab
- Part 2 Volume-matched placebo, intramuscular injection (Placebo Comparator)
  Interventions: Other: Placebo to Biologic

INTERVENTIONS:
Biological: sotrovimab — sotrovimab IV infusion, single dose
  Arms: Part 1 Sotrovimab intravenous infusion, single dose
Other: Placebo to Biologic — Sterile 0.9% (w/v) sodium chloride solution
  Arms: Part 1 Volume-matched placebo, intravenous infusion
Biological: sotrovimab — Sotrovimab IM injection, single dose
  Arms: Part 2 Sotrovimab intramuscular injection, single dose
Other: Placebo to Biologic — Sterile 0.9% (w/v) sodium chloride solution
  Arms: Part 2 Volume-matched placebo, intramuscular injection

SUMMARY:
This is a Phase I single-dose study to investigate the pharmacokinetics, safety, and tolerability of sotrovimab vs placebo by intravenous or intramuscular administration in healthy Japanese and Caucasian participants.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety, tolerability, and pharmacokinetics (PK) of a single fixed dose of sotrovimab administered intravenously (IV) or via intramuscular (IM) injection in Japanese and Caucasian healthy volunteers. This study will occur in two parts (Part 1 and Part 2).

Part 1: Healthy Japanese and Caucasian participants will be randomized in a 4:1 ratio to receive a single IV infusion of sotrovimab or volume-matched saline placebo on Day 1. Participants will be blinded to study intervention. Safety, tolerability, immunogenicity, and PK of IV sotrovimab will be evaluated.

Part 2: Healthy Japanese and Caucasian participants will be randomized in a 4:1 ratio to receive a single IM dose of sotrovimab or volume-matched saline placebo on Day 1. Participants will be blinded to study intervention. Safety, tolerability, immunogenicity, and PK of IM sotrovimab will be evaluated.

The data from this study will be used to supplement data available from other clinical trials that were conducted in non-Japanese participants.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants, aged 18 to 65 years, inclusive
* Participants who are healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring.
* Japanese participants must be of Japanese ancestry, defined as having been born in Japan, being descendants of four ethnic Japanese grandparents and two ethnic Japanese parents, holding a Japanese passport or identity papers, and being able to speak Japanese. Participants should have lived outside Japan for fewer than 10 years at the time of Screening.
* Caucasian participants must be of Caucasian ancestry, defined as Caucasian descent as evidenced by appearance and verbal confirmation of familial heritage.
* Body mass index (BMI) within the range of 18 to 29.9 kg/m2 (inclusive).
* Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the consent form and protocol.

Exclusion Criteria:

* History or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study intervention or interfering with the interpretation of data.
* Lymphoma, leukemia, or any malignancy within the past 5 years except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years.
* Breast cancer within the past 10 years.
* Abnormal blood pressure at Screening.
* Significant allergies to humanized monoclonal antibodies.
* Clinically significant multiple or severe drug allergies, intolerance to topical corticosteroids, or severe post-treatment hypersensitivity reactions (including, but not limited to, erythema multiforme major, linear immunoglobulin A (IgA) dermatosis, toxic epidermal necrolysis, and exfoliative dermatitis).
* Current or chronic history of liver disease or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Use of any prescription medications (besides contraceptive medications or devices) within the 28 days prior to dosing or concomitantly, unless permitted by the protocol or approved by the Investigator in conjunction with the GSK medical monitor.
* Treatment with biologic agents (such as monoclonal antibodies including marketed drugs) within 3 months or 5 half-lives (whichever is longer) prior to dosing.
* Receipt of convalescent plasma from a recovered COVID-19 patient or anti-SARSCoV- 2 mAb within the last 3 months.
* Receipt of any vaccine within 48 hours prior to enrollment. Vaccination will not be allowed for 90 days after dosing.
* Participant has received a SARS-CoV-2 vaccine but has not completed all doses in the series more than 28 days prior to Screening
* Participation in the study would result in loss of blood or blood products in excess of 500 mL within a 56 day period.
* Exposure to more than 4 new chemical entities within 12 months prior to the first dosing day.
* Enrollment in any investigational vaccine study within the last 180 days or any other investigational drug study within 30 days prior to Day 1 or within 5 half-lives of the investigational compound, whichever is longer.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 prior to dosing.
* Positive pre-study drug/alcohol screen.
* Positive HIV antibody test.
* History of regular alcohol consumption within 6 months prior to the study defined as: An average weekly intake of >14 units. One unit is equivalent to 8 g of alcohol: a half pint (~240 mL) of beer, 1 glass (125 mL) of wine, or 1 (25 mL) measure of spirits.
* Regular use of known drugs of abuse.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-07-06 (Actual); Primary Completion 2021-09-02 (Actual); Study Completion 2021-12-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Investigative Site, Anaheim, California
  - Investigative Site, Glendale, California

REFERENCES:
- [Derived] Nader A, Alexander E, Brintziki D, Haggag AZ, Harrison SA, Hawes IA, Hezareh M, Lippa AM, Okamasa A, Okour M, Okuda N, Sager JE, Segal S, Shida Y, Skingsley A, Williams R, Yoon EY, Austin D. Pharmacokinetics, Safety, and Tolerability of Anti-SARS-CoV-2 Monoclonal Antibody, Sotrovimab, Delivered Intravenously or Intramuscularly in Japanese and Caucasian Healthy Volunteers. Clin Pharmacokinet. 2024 Jan;63(1):57-68. doi: 10.1007/s40262-023-01319-2. Epub 2023 Nov 13. PMID 37955825

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in the United States.
Pre-assignment Details: A total of 48 participants (24 participants in Part 1 and 24 participants in Part 2) were enrolled in the study (Safety Population comprised of all randomized participants who were exposed to study intervention).
Groups:
- Part 1: Placebo IV (Japanese): Japanese participants received a volume-matched saline placebo (Sterile 0.9 percent [%] weight/volume [w/v] sodium chloride solution) matching intravenous (IV) infusion of sotrovimab on Day 1.
- Part 1:Placebo IV (Caucasian): Caucasian participants received a volume-matched saline placebo (Sterile 0.9% [w/v] sodium chloride solution) matching IV infusion of sotrovimab on Day 1
- Part 1: Sotrovimab 500 mg IV (Japanese): Japanese participants received a single 500 milligrams (mg) IV infusion of sotrovimab on Day 1
- Part 1: Sotrovimab 500 mg IV (Caucasian): Caucasian participants received a single 500 mg IV infusion of sotrovimab on Day 1
- Part 2: Placebo IM (Japanese): Japanese participants received a volume-matched saline placebo (Sterile 0.9% [w/v] sodium chloride solution) matching intramuscular (IM) injection of sotrovimab on Day 1.
- Part 2: Placebo IM (Caucasian): Caucasian participants received a volume-matched saline placebo (Sterile 0.9% [w/v] sodium chloride solution) matching IM injection of sotrovimab on Day 1.
- Part 2: Sotrovimab 500 mg IM (Japanese): Japanese participants received a single 500 mg IM injection of sotrovimab (administered as two 4 milliliters [mL] injections, one in each dorsogluteal muscle) on Day 1.
- Part 2: Sotrovimab 500 mg IM (Caucasian): Caucasian participants received a single 500 mg IM injection of sotrovimab (administered as two 4 mL injections, one in each dorsogluteal muscle) on Day 1.
Period: Part 1 (Up to Week 18)
Arm/Group | Part 1: Placebo IV (Japanese) | Part 1:Placebo IV (Caucasian) | Part 1: Sotrovimab 500 mg IV (Japanese) | Part 1: Sotrovimab 500 mg IV (Caucasian) | Part 2: Placebo IM (Japanese) | Part 2: Placebo IM (Caucasian) | Part 2: Sotrovimab 500 mg IM (Japanese) | Part 2: Sotrovimab 500 mg IM (Caucasian)
Started | 3 | 3 | 9 | 9 | 0 | 0 | 0 | 0
Completed | 3 | 3 | 9 | 9 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2 (Up to Week 18)
Arm/Group | Part 1: Placebo IV (Japanese) | Part 1:Placebo IV (Caucasian) | Part 1: Sotrovimab 500 mg IV (Japanese) | Part 1: Sotrovimab 500 mg IV (Caucasian) | Part 2: Placebo IM (Japanese) | Part 2: Placebo IM (Caucasian) | Part 2: Sotrovimab 500 mg IM (Japanese) | Part 2: Sotrovimab 500 mg IM (Caucasian)
Started | 0 | 0 | 0 | 0 | 2 | 2 | 10 | 10
Completed | 0 | 0 | 0 | 0 | 2 | 2 | 10 | 10
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were reported for the Safety Population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: Placebo IV (Japanese) | Part 1:Placebo IV (Caucasian) | Part 1: Sotrovimab 500 mg IV (Japanese) | Part 1: Sotrovimab 500 mg IV (Caucasian) | Part 2: Placebo IM (Japanese) | Part 2: Placebo IM (Caucasian) | Part 2: Sotrovimab 500 mg IM (Japanese) | Part 2: Sotrovimab 500 mg IM (Caucasian) | Total
Number analyzed (Participants) | 3 | 3 | 9 | 9 | 2 | 2 | 10 | 10 | 48
Age, Customized [Count of Participants; unit: Participants]
  Participants: <=18 Years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Participants: 19-64 Years | 3 | 3 | 9 | 9 | 2 | 2 | 10 | 10 | 48
  Participants: >=65 Years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 8 | 5 | 2 | 1 | 7 | 7 | 33
  Male | 1 | 2 | 1 | 4 | 0 | 1 | 3 | 3 | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Participants: ASIAN-JAPANESE HERITAGE | 3 | 0 | 9 | 0 | 2 | 0 | 10 | 0 | 24
  Participants: WHITE-WHITE/CAUCASIAN/EUROPEAN HERITAGE | 0 | 3 | 0 | 9 | 0 | 2 | 0 | 10 | 24

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Maximum Observed Serum Concentration (Cmax) of Sotrovimab Through Day 29
Description: The Cmax was summarized using standard non-compartmental pharmacokinetic analysis methods. The geometric means and geometric coefficient of variation are presented. An ethnicity comparison (Japanese versus Caucasian) was also conducted using analysis of covariance (ANCOVA) adjusting for body weight. The geometric Least Square (LS) means ratio (Japanese versus Caucasian) for Cmax and 90 percent (%) confidence interval (CI) are presented.
Time Frame: Day 1: Pre-dose, at end of infusion (EOI) and 1, 2, 6, 8, 24 (Day 2) and 48 (Day 3) hours after end of infusion; Days 8, 15 and 29
Population: Pharmacokinetic Population comprised all participants in the Safety Population (All randomized participants who were exposed to study intervention) who had at least 1 non-missing PK assessment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | Part 1: Sotrovimab 500 mg IV (Japanese) | Part 1: Sotrovimab 500 mg IV (Caucasian)
Number analyzed (Participants) | 9 | 9
Micrograms per milliliter | 238.32 (18.5) | 188.66 (13.8)
Statistical Analysis 1: Comparison: Part 1: Sotrovimab 500 mg IV (Japanese) vs Part 1: Sotrovimab 500 mg IV (Caucasian); Test type: Superiority; Ratio of geometric least squares means = 1.0724, 90% CI 2-sided [0.8519 to 1.3500] — The ratio of geometric LS means and 90% confidence intervals were obtained from ANCOVA model, with Cmax as the dependent variable, and ethnicity and body weight were covariates

2. Primary Outcome: Part 1: Area Under the Serum-concentration Time Curve From Day 1 to Day 29 (AUC[D1-29]) of Sotrovimab
Description: The AUC (D1-29) was summarized using standard non-compartmental pharmacokinetic analysis methods. The geometric mean and geometric coefficient of variation are presented. An ethnicity comparison (Japanese versus Caucasian) was also conducted using ANCOVA adjusting for body weight. The geometric LS means ratio (Japanese versus Caucasian) for AUC(D1-29) and 90% Confidence Interval are presented.
Time Frame: Day 1: Pre-dose, at end of infusion and 1, 2, 6, 8, 24 (Day 2) and 48 (Day 3) hours after end of infusion; Days 8, 15 and 29
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Day*micrograms per milliliter
Arm/Group | Part 1: Sotrovimab 500 mg IV (Japanese) | Part 1: Sotrovimab 500 mg IV (Caucasian)
Number analyzed (Participants) | 9 | 9
Day*micrograms per milliliter | 2699.29 (11.5) | 2154.90 (9.0)
Statistical Analysis 1: Comparison: Part 1: Sotrovimab 500 mg IV (Japanese) vs Part 1: Sotrovimab 500 mg IV (Caucasian); Test type: Other; Ratio of geometric least squares means = 1.0513, 90% CI 2-sided [0.9281 to 1.1908] — The ratio of geometric LS means and 90% confidence intervals were obtained from ANCOVA model, with AUC(D1-29) as the dependent variable, and ethnicity and body weight were covariates

3. Primary Outcome: Part 1: Time to Cmax (Tmax) of Sotrovimab Through Day 29
Description: The Tmax was summarized using standard non-compartmental pharmacokinetic analysis methods. The median and full range are presented.
Time Frame: as for outcome 2
Population: Pharmacokinetic Population. Only those participants with data available at specified time point were analyzed. Participants with slow drug distribution following IV infusion were excluded.
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1: Sotrovimab 500 mg IV (Japanese) | Part 1: Sotrovimab 500 mg IV (Caucasian)
Number analyzed (Participants) | 9 | 8
Hours | 1.567 [1.55 to 6.55] | 0.733 [0.68 to 1.58]

4. Primary Outcome: Part 1: Concentration at Day 29 (CD29) Following Administration of Sotrovimab
Description: The CD29 was summarized using standard non-compartmental pharmacokinetic analysis methods. The geometric mean and geometric coefficient of variation are presented.
Time Frame: as for outcome 2
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | Part 1: Sotrovimab 500 mg IV (Japanese) | Part 1: Sotrovimab 500 mg IV (Caucasian)
Number analyzed (Participants) | 9 | 9
Micrograms per milliliter | 71.48 (15.1) | 55.56 (9.1)

5. Primary Outcome: Part 2: Cmax of Sotrovimab Through Day 29
Description: The Cmax was summarized using standard non-compartmental pharmacokinetic analysis methods. The geometric mean and geometric coefficient of variation are presented. An ethnicity comparison (Japanese versus Caucasian) was also conducted using ANCOVA adjusting for body weight. The geometric LS means ratio (Japanese versus Caucasian) for Cmax and 90% confidence interval are presented.
Time Frame: Day 1: Pre-dose and 1, 2, 6, 8, 24 (Day 2) and 48 (Day 3) hours after first IM injection; Days 8, 15 and 29
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | Part 2: Sotrovimab 500 mg IM (Japanese) | Part 2: Sotrovimab 500 mg IM (Caucasian)
Number analyzed (Participants) | 10 | 10
Micrograms per milliliter | 60.33 (32.0) | 32.27 (50.4)
Statistical Analysis 1: Comparison: Part 2: Sotrovimab 500 mg IM (Japanese) vs Part 2: Sotrovimab 500 mg IM (Caucasian); Test type: Other; Ratio of geometric least squares means = 1.6999, 90% CI 2-sided [1.1500 to 2.5129] — [estimate comment as in outcome 1, analysis 1]

6. Primary Outcome: Part 2: AUC(D1-29) of Sotrovimab
Description: as for outcome 2
Time Frame: Day 1: Pre-dose and 1, 2, 6, 8, 24 (Day 2) and 48 (Day 3) hours after first IM injection; Days 8, 15 and 29
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Day*micrograms per milliliter
Arm/Group | Part 2: Sotrovimab 500 mg IM (Japanese) | Part 2: Sotrovimab 500 mg IM (Caucasian)
Number analyzed (Participants) | 10 | 10
Day*micrograms per milliliter | 1378.28 (28.1) | 743.39 (46.4)
Statistical Analysis 1: Comparison: Part 2: Sotrovimab 500 mg IM (Japanese) vs Part 2: Sotrovimab 500 mg IM (Caucasian); Test type: Other; Ratio of geometric least squares means = 1.5869, 90% CI 2-sided [1.1236 to 2.2413] — [estimate comment as in outcome 2, analysis 1]

7. Primary Outcome: Part 2: Tmax of Sotrovimab Through Day 29
Description: as for outcome 3
Time Frame: Day 1: Pre-dose and 1, 2, 6, 8, 24 (Day 2) and 48 (Day 3) hours after first IM injection; Days 8, 15 and 29
Population: Pharmacokinetic Population
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 2: Sotrovimab 500 mg IM (Japanese) | Part 2: Sotrovimab 500 mg IM (Caucasian)
Number analyzed (Participants) | 10 | 10
Hours | 168.88 [167.8 to 334.1] | 166.60 [165.4 to 696.4]

8. Primary Outcome: Part 2: CD29 of Sotrovimab
Description: as for outcome 4
Time Frame: Day 1: Pre-dose and 1, 2, 6, 8, 24 (Day 2) and 48 (Day 3) hours after first IM injection; Days 8, 15 and 29
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | Part 2: Sotrovimab 500 mg IM (Japanese) | Part 2: Sotrovimab 500 mg IM (Caucasian)
Number analyzed (Participants) | 10 | 10
Micrograms per milliliter | 44.5 (30.5) | 29.14 (50.9)

9. Primary Outcome: Part 1: Number of Participants With Serious Adverse Events (SAE) and Common Non-serious Adverse Events (Non-SAE) Through Day 29
Description: An adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. An SAE is defined as any serious adverse event that, at any dose: results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or any other situations as per medical or scientific judgment. Adverse events which were not serious adverse events were considered as Non-Serious adverse events.
Time Frame: Up to Day 29
Population: Safety Population comprised of all randomized participants who were exposed to study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Placebo IV (Japanese) | Part 1:Placebo IV (Caucasian) | Part 1: Sotrovimab 500 mg IV (Japanese) | Part 1: Sotrovimab 500 mg IV (Caucasian)
Number analyzed (Participants) | 3 | 3 | 9 | 9
Participants
  SAE | 0 | 0 | 0 | 0
  Non-SAE | 1 | 1 | 2 | 1

10. Primary Outcome: Part 1: Number of Participants With Adverse Events of Special Interest (AESI) Through Day 29
Description: Adverse events of special interest (AESI) are relevant known toxicities of other therapeutic monoclonal antibodies (mAbs) or signals observed in nonclinical programs of sotrovimab. AESI were defined as Infusion-related reactions (IRR) including hypersensitivity reactions, Hypersensitivity Standardized Medical dictionary for Regulatory Activities (MedDRA) Queries (SMQ) narrow, Infusion site reactions, Immunogenicity related adverse drug reactions (ADR) and AE potentially related to antibody-dependent enhancement of disease (ADE). Only IRR including hypersensitivity and Infusion site reactions through Day 29 were summarized.
Time Frame: Up to Day 29
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Placebo IV (Japanese) | Part 1:Placebo IV (Caucasian) | Part 1: Sotrovimab 500 mg IV (Japanese) | Part 1: Sotrovimab 500 mg IV (Caucasian)
Number analyzed (Participants) | 3 | 3 | 9 | 9
Participants
  IRR including hypersensitivity | 0 | 0 | 0 | 0
  Infusion Site Reactions | 0 | 0 | 0 | 0

11. Primary Outcome: Part 1: Number of Participants With Abnormal Clinically Significant Electrocardiogram (ECG) Findings Through Day 29
Description: Twelve-lead ECG's were obtained in the semi-recumbent or supine position after 10 minutes of rest using an ECG machine. Clinically significant abnormal findings are those which are not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition. Data for the number of participants with abnormal clinically significant worst case post-Baseline ECG findings were reported.
Time Frame: Up to Day 29
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Placebo IV (Japanese) | Part 1:Placebo IV (Caucasian) | Part 1: Sotrovimab 500 mg IV (Japanese) | Part 1: Sotrovimab 500 mg IV (Caucasian)
Number analyzed (Participants) | 3 | 3 | 9 | 9
Participants | 0 | 0 | 0 | 0

12. Primary Outcome: Part 1: Number of Participants With Vital Signs Grade Shifts From Baseline Grade Through Day 29
Description: Vital signs including systolic blood pressure (SBP), diastolic blood pressure (DBP) and pulse rate were measured in a semi-supine or sitting position after 5 minutes rest. Baseline is latest pre-dose assessment with a non-missing value on or after Day -1 visit including those from unscheduled visits. Grade Shift from Baseline is defined as shift from any grade (at Baseline) to Grades 1, 2, 3 and 4 post-Baseline. A worst post-Baseline grade shift is defined as worst change that occurred at any measured time point during treatment period. Grading was determined by the Division of Acquired Immunodeficiency Syndrome Table for Grading Severity (DAIDS) version 2.1. Grade 0=Normal, Grade 1=Mild, Grade 2=Moderate, Grade 3=Severe and Grade 4= Potentially Life-Threatening. Data is presented for only those parameters for which participants had grade shifts from Baseline grade. Worst-case post-Baseline shift data is presented.
Time Frame: Baseline (Day 1) and up to Day 29
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Placebo IV (Japanese) | Part 1:Placebo IV (Caucasian) | Part 1: Sotrovimab 500 mg IV (Japanese) | Part 1: Sotrovimab 500 mg IV (Caucasian)
Number analyzed (Participants) | 3 | 3 | 9 | 9
Participants | 0 | 0 | 0 | 0

13. Primary Outcome: Part 1: Number of Participants With Clinical Chemistry Grade Shifts From Baseline Grade Through Day 29
Description: Blood samples were collected for analysis of clinical chemistry parameters including Total Bilirubin, Direct Bilirubin, Glucose (fasting) and Glucose. Baseline is latest pre-dose assessment with a non-missing value on or after Day -1 visit including those from unscheduled visits. Grade Shift from Baseline is defined as shift from any grade (at Baseline) to Grades 1, 2, 3 and 4 post-Baseline. A worst post-Baseline grade shift is defined as worst change that occurred at any measured time point during treatment period. Grading was determined by the Division of Acquired Immunodeficiency Syndrome (AIDS) Table for Grading Severity (DAIDS) version 2.1. Grade 0=Normal, Grade 1=Mild, Grade 2=Moderate, Grade 3=Severe and Grade 4= Potentially Life-Threatening. Data is presented for only those parameters for which participants had grade shifts from Baseline grade. Worst-case post-Baseline shift data is presented.
Time Frame: Baseline (Day 1) and up to Day 29
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Placebo IV (Japanese) | Part 1:Placebo IV (Caucasian) | Part 1: Sotrovimab 500 mg IV (Japanese) | Part 1: Sotrovimab 500 mg IV (Caucasian)
Number analyzed (Participants) | 3 | 3 | 9 | 9
Participants
  Total Bilirubin, High, Grade 0 to Grade 1 | 0 | 1 | 1 | 0
  Direct Bilirubin, High, Grade 0 to Grade 3 | 0 | 0 | 1 | 0
  Glucose (fasting), High, Grade 0 to Grade 1 | 0 | 0 | 0 | 2
  Glucose (fasting), High, Grade 0 to Grade 2 | 0 | 0 | 0 | 1
  Glucose, Low, Grade 1 to Grade 0 | 0 | 1 | 0 | 0

14. Primary Outcome: Part 1: Number of Participants With Any Increase in Worst-case Urinalysis Results Post-Baseline Relative to Baseline by Dipstick Method Through Day 29
Description: Urine samples were collected for analysis of bilirubin, leukocyte esterase, occult blood, and protein by a dipstick method. The dipstick test gives results in a semi-quantitative manner indicating proportional concentrations in the urine sample. Baseline is defined as the latest pre-dose assessment with a non-missing value on or after Day -1 visit, including those from unscheduled visits. Any increase means any increase to small, moderate, severe, potentially life threatening or positive post-Baseline relative to Baseline. Data is presented for only those parameters for which participants had any increase in urinalysis results post-Baseline relative to Baseline. Number of participants with worst case any increase in urinalysis results post-Baseline relative to Baseline has been presented.
Time Frame: Baseline (Day 1) and up to Day 29
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Placebo IV (Japanese) | Part 1:Placebo IV (Caucasian) | Part 1: Sotrovimab 500 mg IV (Japanese) | Part 1: Sotrovimab 500 mg IV (Caucasian)
Number analyzed (Participants) | 3 | 3 | 9 | 9
Participants
  Bilirubin | 1 | 0 | 2 | 0
  Leukocyte Esterase | 0 | 0 | 2 | 0
  Occult Blood | 0 | 0 | 3 | 2
  Protein | 0 | 0 | 1 | 0

15. Primary Outcome: Part 2: Number of Participants With SAE and Common Non-SAE Through Day 29
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. An SAE is defined as any serious adverse event that, at any dose, results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or any other situations as per medical or scientific judgment. Adverse events which were not serious adverse events were considered as Non-Serious adverse events.
Time Frame: Part 2: Number of participants with SAE and common non-SAE through Day 29
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Placebo IM (Japanese) | Part 2: Placebo IM (Caucasian) | Part 2: Sotrovimab 500 mg IM (Japanese) | Part 2: Sotrovimab 500 mg IM (Caucasian)
Number analyzed (Participants) | 2 | 2 | 10 | 10
Participants
  SAE | 0 | 0 | 0 | 0
  Non-SAE | 0 | 1 | 4 | 2

16. Primary Outcome: Part 2: Number of Participants With AESI Through Day 29
Description: Adverse events of special interest (AESI) are relevant known toxicities of other therapeutic mAbs or signals observed in nonclinical programs of sotrovimab. AESI were defined as Injection-related reactions including hypersensitivity reactions, Hypersensitivity (SMQ narrow), Injection site reactions, Immunogenicity related adverse drug reactions (ADR) and AE potentially related to antibody-dependent enhancement of disease (ADE). Only Injection-related reactions including hypersensitivity and Injection site reactions through Day 29 were summarized.
Time Frame: Up to Day 29
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Placebo IM (Japanese) | Part 2: Placebo IM (Caucasian) | Part 2: Sotrovimab 500 mg IM (Japanese) | Part 2: Sotrovimab 500 mg IM (Caucasian)
Number analyzed (Participants) | 2 | 2 | 10 | 10
Participants
  Injection-related reactions including hypersensitivity | 0 | 0 | 0 | 0
  Injection Site Reaction | 0 | 0 | 1 | 0

17. Primary Outcome: Part 2: Number of Participants With Abnormal Clinically Significant ECG Findings Through Day 29
Description: as for outcome 11
Time Frame: Up to Day 29
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Placebo IM (Japanese) | Part 2: Placebo IM (Caucasian) | Part 2: Sotrovimab 500 mg IM (Japanese) | Part 2: Sotrovimab 500 mg IM (Caucasian)
Number analyzed (Participants) | 2 | 2 | 10 | 10
Participants | 0 | 0 | 0 | 0

18. Primary Outcome: Part 2: Number of Participants With Vital Signs Grade Shifts From Baseline Grade Through Day 29
Description: Vital signs including SBP, DBP and pulse rate were measured in a semi-supine or sitting position after 5 minutes rest. Baseline is latest pre-dose assessment with a non-missing value on or after Day -1 visit including those from unscheduled visits. Grade Shift from Baseline is defined as shift from any grade (at Baseline) to Grades 1, 2, 3 and 4 post-Baseline. A worst post-Baseline grade shift is defined as worst change that occurred at any measured time point during treatment period. Grading was determined by the Division of Acquired Immunodeficiency Syndrome Table for Grading Severity (DAIDS) version 2.1. Grade 0=Normal, Grade 1=Mild, Grade 2=Moderate, Grade 3=Severe and Grade 4= Potentially Life-Threatening. Worst-case post-Baseline shift data is presented.
Time Frame: Baseline (Day) and up to Day 29
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Placebo IM (Japanese) | Part 2: Placebo IM (Caucasian) | Part 2: Sotrovimab 500 mg IM (Japanese) | Part 2: Sotrovimab 500 mg IM (Caucasian)
Number analyzed (Participants) | 2 | 2 | 10 | 10
Participants
  DBP; Grade 0 to Grade 1 | 0 | 0 | 0 | 0
  SBP; Grade 1 to Grade 0 | 0 | 0 | 1 | 0
  Pulse rate; Grade 0 to Grade 1 | 0 | 0 | 0 | 0

19. Primary Outcome: Part 2: Number of Participants With Clinical Chemistry Grade Shifts From Baseline Grade Through Day 29
Description: Blood samples were collected for analysis of clinical chemistry parameters including Alkaline Phosphatase (ALP), Total Bilirubin, Glucose, Potassium and Sodium. Baseline is latest pre-dose assessment with a non-missing value on or after Day -1 visit including those from unscheduled visits. Grade Shift from Baseline is defined as shift from any grade (at Baseline) to Grades 1, 2, 3 and 4 post-Baseline. A worst post-Baseline grade shift is defined as worst change that occurred at any measured time point during treatment period. Grading was determined by the Division of Acquired Immunodeficiency Syndrome (AIDS) Table for Grading Severity (DAIDS) version 2.1. Grade 0=Normal, Grade 1=Mild, Grade 2=Moderate, Grade 3=Severe and Grade 4= Potentially Life-Threatening. Data is presented for only those parameters for which participants had grade shifts from Baseline grade. Worst-case post-Baseline shift data is presented.
Time Frame: Baseline (Day 1) and up to Day 29
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Placebo IM (Japanese) | Part 2: Placebo IM (Caucasian) | Part 2: Sotrovimab 500 mg IM (Japanese) | Part 2: Sotrovimab 500 mg IM (Caucasian)
Number analyzed (Participants) | 2 | 2 | 10 | 10
Participants
  ALP, High, Grade 0 to Grade 1 | 0 | 0 | 0 | 1
  Total Bilirubin, High, Grade 0 to Grade 1 | 0 | 0 | 1 | 0
  Glucose, Low, Grade 0 to Grade 1 | 1 | 0 | 0 | 0
  Potassium, High, Grade 0 to Grade 4 | 0 | 0 | 1 | 0
  Sodium, Low, Grade 1 to Grade 1 | 0 | 0 | 1 | 1

20. Primary Outcome: Part 2: Number of Participants With Any Increase in Worst-case Urinalysis Results Post-Baseline Relative to Baseline by Dipstick Method Through Day 29
Description: Urine samples were collected for analysis of bilirubin, glucose, leukocyte esterase, occult blood and protein by a dipstick method. The dipstick test gives results in a semi-quantitative manner indicating proportional concentrations in the urine sample. Baseline is defined as the latest pre-dose assessment with a non-missing value on or after Day -1 visit, including those from unscheduled visits. Any increase means any increase to small, moderate, severe, potentially life threatening or positive post-Baseline relative to Baseline. Data is presented for only those parameters for which participants had any increase in urinalysis results post-Baseline relative to Baseline. Number of participants with worst case any increase in urinalysis results post-Baseline relative to Baseline has been presented.
Time Frame: Baseline (Day 1) and up to Day 29
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Placebo IM (Japanese) | Part 2: Placebo IM (Caucasian) | Part 2: Sotrovimab 500 mg IM (Japanese) | Part 2: Sotrovimab 500 mg IM (Caucasian)
Number analyzed (Participants) | 2 | 2 | 10 | 10
Participants
  Bilirubin | 1 | 0 | 0 | 0
  Glucose | 0 | 0 | 1 | 0
  Leukocyte Esterase | 0 | 0 | 1 | 2
  Occult Blood | 1 | 1 | 1 | 4
  Protein | 0 | 0 | 1 | 2

21. Secondary Outcome: Part 1: Cmax of Sotrovimab Through Week 18
Description: as for outcome 5
Time Frame: Day 1: Pre-dose, at end of infusion and 1, 2, 6, 8, 24 (Day 2) and 48 (Day 3) hours after end of infusion; Weeks 2, 3, 4, 6, 8, 12 and 18
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | Part 1: Sotrovimab 500 mg IV (Japanese) | Part 1: Sotrovimab 500 mg IV (Caucasian)
Number analyzed (Participants) | 9 | 9
Micrograms per milliliter | 238.32 (18.5) | 188.66 (13.8)
Statistical Analysis 1: Comparison: Part 1: Sotrovimab 500 mg IV (Japanese) vs Part 1: Sotrovimab 500 mg IV (Caucasian); Test type: Other; Ratio of geometric least squares means = 1.0724, 90% CI 2-sided [0.8519 to 1.3500] — [estimate comment as in outcome 1, analysis 1]

22. Secondary Outcome: Part 1: Area Under the Serum Concentration-time Curve Extrapolated to Infinite Time (AUC[0-infinity]) of Sotrovimab Through Week 18
Description: The AUC(0-infinity) was summarized using standard non-compartmental pharmacokinetic analysis methods. The geometric mean and geometric coefficient of variation are presented.
Time Frame: as for outcome 21
Population: Pharmacokinetic Population. Only those participants with data available at specified time points were analyzed. Participants with the extrapolated portion of AUCinfinity (% AUCex) >20% were excluded.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Day*micrograms per milliliter
Arm/Group | Part 1: Sotrovimab 500 mg IV (Japanese) | Part 1: Sotrovimab 500 mg IV (Caucasian)
Number analyzed (Participants) | 3 | 2
Day*micrograms per milliliter | 7513.23 (22.1) | 5388.17 (30.8)

23. Secondary Outcome: Part 1: Area Under the Curve From the Time of Dosing to the Time of the Last Measurable (Positive) Concentration (AUClast) of Sotrovimab Through Week 18
Description: The AUClast was summarized using standard non-compartmental pharmacokinetic analysis methods. The geometric mean and geometric coefficient of variation are presented. An ethnicity comparison (Japanese versus Caucasian) was also conducted using ANCOVA adjusting for body weight. The geometric LS means ratio (Japanese versus Caucasian) for AUClast and 90% Confidence Interval are presented.
Time Frame: as for outcome 21
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Day*micrograms per milliliter
Arm/Group | Part 1: Sotrovimab 500 mg IV (Japanese) | Part 1: Sotrovimab 500 mg IV (Caucasian)
Number analyzed (Participants) | 9 | 9
Day*micrograms per milliliter | 6597.35 (10.9) | 5098.64 (12.0)
Statistical Analysis 1: Comparison: Part 1: Sotrovimab 500 mg IV (Japanese) vs Part 1: Sotrovimab 500 mg IV (Caucasian); Test type: Other; Ratio of geometric least squares means = 1.0673, 90% CI 2-sided [0.9286 to 1.2268] — The ratio of geometric LS means and 90% confidence intervals were obtained from ANCOVA model, with AUClast as the dependent variable, and ethnicity and body weight were covariates

24. Secondary Outcome: Part 1: Tmax of Sotrovimab Through Week 18
Description: as for outcome 3
Time Frame: as for outcome 21
Population: Pharmacokinetic Population. Only those participants with data available at specified time points were analyzed. Participants with slow drug distribution following IV infusion were excluded.
Measure: Median (Full Range); unit: Day
Arm/Group | Part 1: Sotrovimab 500 mg IV (Japanese) | Part 1: Sotrovimab 500 mg IV (Caucasian)
Number analyzed (Participants) | 9 | 8
Day | 0.065 [0.06 to 0.27] | 0.031 [0.03 to 0.07]

25. Secondary Outcome: Part 1: Time of the Last Quantifiable Concentration (Tlast) of Sotrovimab Through Week 18
Description: The Tlast was summarized using standard non-compartmental pharmacokinetic analysis methods. The median and full range are presented.
Time Frame: as for outcome 21
Population: Pharmacokinetic Population
Measure: Median (Full Range); unit: Day
Arm/Group | Part 1: Sotrovimab 500 mg IV (Japanese) | Part 1: Sotrovimab 500 mg IV (Caucasian)
Number analyzed (Participants) | 9 | 9
Day | 125.98 [119.0 to 126.1] | 125.98 [125.0 to 127.1]

26. Secondary Outcome: Part 1: Terminal Elimination Half-life (t1/2) of Sotrovimab Through Week 18
Description: The T1/2 was summarized using standard non-compartmental pharmacokinetic analysis methods. The median and full range are presented.
Time Frame: Weeks 2, 3, 4, 6, 8, 12 and 18
Population: Pharmacokinetic Population
Measure: Median (Full Range); unit: Day
Arm/Group | Part 1: Sotrovimab 500 mg IV (Japanese) | Part 1: Sotrovimab 500 mg IV (Caucasian)
Number analyzed (Participants) | 9 | 9
Day | 56.38 [40.9 to 65.7] | 58.85 [33.6 to 113.6]

27. Secondary Outcome: Part 2: Cmax of Sotrovimab Through Week 18
Description: as for outcome 5
Time Frame: Day 1: Pre-dose and 1, 2, 6, 8, 24 (Day 2) and 48 (Day 3) hours after first IM injection; Weeks 2, 3, 4, 6, 8, 12 and 18
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | Part 2: Sotrovimab 500 mg IM (Japanese) | Part 2: Sotrovimab 500 mg IM (Caucasian)
Number analyzed (Participants) | 10 | 10
Micrograms per milliliter | 60.33 (32.0) | 32.27 (50.4)
Statistical Analysis 1: Comparison: Part 2: Sotrovimab 500 mg IM (Japanese) vs Part 2: Sotrovimab 500 mg IM (Caucasian); Test type: Other; Ratio of geometric least squares means = 1.6999, 90% CI 2-sided [1.1500 to 2.5129] — [estimate comment as in outcome 1, analysis 1]

28. Secondary Outcome: Part 2: AUC(0-infinity) of Sotrovimab Through Week 18
Description: The AUC0-infinity was summarized using standard non-compartmental pharmacokinetic analysis methods. The geometric mean and geometric coefficient of variation are presented.
Time Frame: as for outcome 27
Population: as for outcome 22
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Day*micrograms per milliliter
Arm/Group | Part 2: Sotrovimab 500 mg IM (Japanese) | Part 2: Sotrovimab 500 mg IM (Caucasian)
Number analyzed (Participants) | 1 | 2
Day*micrograms per milliliter | 5687.48 (NA) — NA indicates that data was not available as geometric coefficient of variation could not be calculated for a single participant. | 2788.57 (60.9)

29. Secondary Outcome: Part 2: AUClast of Sotrovimab Through Week 18
Description: as for outcome 23
Time Frame: as for outcome 27
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Day*micrograms per milliliter
Arm/Group | Part 2: Sotrovimab 500 mg IM (Japanese) | Part 2: Sotrovimab 500 mg IM (Caucasian)
Number analyzed (Participants) | 10 | 10
Day*micrograms per milliliter | 4018.36 (25.1) | 2148.93 (39.6)
Statistical Analysis 1: Comparison: Part 2: Sotrovimab 500 mg IM (Japanese) vs Part 2: Sotrovimab 500 mg IM (Caucasian); Test type: Other; Ratio of geometric least squares means = 1.5766, 90% CI 2-sided [1.1777 to 2.1106] — [estimate comment as in outcome 23, analysis 1]

30. Secondary Outcome: Part 2: Tmax of Sotrovimab Through Week 18
Description: as for outcome 3
Time Frame: as for outcome 27
Population: Pharmacokinetic Population
Measure: Median (Full Range); unit: Day
Arm/Group | Part 2: Sotrovimab 500 mg IM (Japanese) | Part 2: Sotrovimab 500 mg IM (Caucasian)
Number analyzed (Participants) | 10 | 10
Day | 7.04 [7.0 to 13.9] | 6.94 [6.9 to 29.0]

31. Secondary Outcome: Part 2: Tlast of Sotrovimab Through Week 18
Description: as for outcome 25
Time Frame: as for outcome 27
Population: Pharmacokinetic Population
Measure: Median (Full Range); unit: Day
Arm/Group | Part 2: Sotrovimab 500 mg IM (Japanese) | Part 2: Sotrovimab 500 mg IM (Caucasian)
Number analyzed (Participants) | 10 | 10
Day | 127.54 [125.9 to 129.0] | 125.52 [118.9 to 132.0]

32. Secondary Outcome: Part 2: T1/2 of Sotrovimab Through Week 18
Description: as for outcome 26
Time Frame: Weeks 2, 3, 4, 6, 8, 12 and 18
Population: Pharmacokinetic Population. Only those participants with data available at specified time points were analyzed. Participants with adjusted regression coefficient for the slope of elimination phase (R^2) <0.8 were excluded.
Measure: Median (Full Range); unit: Day
Arm/Group | Part 2: Sotrovimab 500 mg IM (Japanese) | Part 2: Sotrovimab 500 mg IM (Caucasian)
Number analyzed (Participants) | 10 | 9
Day | 67.28 [53.2 to 85.5] | 67.40 [48.6 to 89.2]

33. Secondary Outcome: Part 1: Number of Participants With SAE and Common Non-SAE Through Week 18
Description: as for outcome 15
Time Frame: Up to Week 18
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Placebo IV (Japanese) | Part 1:Placebo IV (Caucasian) | Part 1: Sotrovimab 500 mg IV (Japanese) | Part 1: Sotrovimab 500 mg IV (Caucasian)
Number analyzed (Participants) | 3 | 3 | 9 | 9
Participants
  SAE | 0 | 0 | 0 | 0
  Non-SAE | 1 | 1 | 2 | 1

34. Secondary Outcome: Part 1: Number of Participants With AESI Through Week 18
Description: Adverse events of special interest (AESI) are relevant known toxicities of other therapeutic mAbs or signals observed in nonclinical programs of sotrovimab. AESI were defined as Infusion-related reactions (IRR) including hypersensitivity reactions, Hypersensitivity (SMQ narrow), Infusion site reactions, Immunogenicity related adverse drug reactions (ADR) and AE potentially related to antibody-dependent enhancement of disease (ADE).
Time Frame: Up to Week 18
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Placebo IV (Japanese) | Part 1:Placebo IV (Caucasian) | Part 1: Sotrovimab 500 mg IV (Japanese) | Part 1: Sotrovimab 500 mg IV (Caucasian)
Number analyzed (Participants) | 3 | 3 | 9 | 9
Participants
  IRR including hypersensitivity | 0 | 0 | 0 | 0
  Hypersensitivity (SMQ narrow) | 0 | 0 | 1 | 0
  Infusion Site Reaction | 0 | 0 | 0 | 0
  Immunogenicity related ADR | 0 | 0 | 0 | 0
  AE potentially related to ADE | 0 | 0 | 0 | 0

35. Secondary Outcome: Part 1: Number of Participants With Abnormal Clinically Significant ECG Findings Through Week 18
Description: as for outcome 11
Time Frame: Up to Week 18
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Placebo IV (Japanese) | Part 1:Placebo IV (Caucasian) | Part 1: Sotrovimab 500 mg IV (Japanese) | Part 1: Sotrovimab 500 mg IV (Caucasian)
Number analyzed (Participants) | 3 | 3 | 9 | 9
Participants | 0 | 0 | 0 | 0

36. Secondary Outcome: Part 1: Number of Participants With Vital Signs Grade Shifts From Baseline Grade Through Week 18
Description: Vital signs including SBP, DBP and pulse rate were measured in a semi-supine or sitting position after 5 minutes rest. Baseline is latest pre-dose assessment with a non-missing value on or after Day -1 visit including those from unscheduled visits. Grade Shift from Baseline is defined as shift from any grade (at Baseline) to Grades 1, 2, 3 and 4 post-Baseline. A worst post-Baseline grade shift is defined as worst change that occurred at any measured time point during treatment period. Grading was determined by the Division of Acquired Immunodeficiency Syndrome Table for Grading Severity (DAIDS) version 2.1. Grade 0=Normal, Grade 1=Mild, Grade 2=Moderate, Grade 3=Severe and Grade 4= Potentially Life-Threatening. Data is presented for only those parameters for which participants had grade shifts from Baseline grade. Worst-case post-Baseline shift data is presented.
Time Frame: Baseline (Day 1) and up to Week 18
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Placebo IV (Japanese) | Part 1:Placebo IV (Caucasian) | Part 1: Sotrovimab 500 mg IV (Japanese) | Part 1: Sotrovimab 500 mg IV (Caucasian)
Number analyzed (Participants) | 3 | 3 | 9 | 9
Participants | 0 | 0 | 0 | 0

37. Secondary Outcome: Part 1: Number of Participants With Clinical Chemistry Shifts From Baseline Grade Through Week 18
Description: Blood samples were collected for analysis of clinical chemistry parameters including Aspartate Aminotransferase (AST), Total Bilirubin, Direct Bilirubin, Glucose (fasting), Glucose and Sodium. Baseline is latest pre-dose assessment with a non-missing value on or after Day -1 visit including those from unscheduled visits. Grade Shift from Baseline is defined as shift from any grade (at Baseline) to Grades 1, 2, 3 and 4 post-Baseline. A worst post-Baseline grade shift is defined as worst change that occurred at any measured time point during treatment period. Grading was determined by the Division of Acquired Immunodeficiency Syndrome (AIDS) Table for Grading Severity (DAIDS) version 2.1. Grade 0=Normal, Grade 1=Mild, Grade 2=Moderate, Grade 3=Severe and Grade 4= Potentially Life-Threatening. Data is presented for only those parameters for which participants had grade shifts from Baseline grade. Worst-case post-Baseline shift data is presented.
Time Frame: Baseline (Day 1) and up to Week 18
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Placebo IV (Japanese) | Part 1:Placebo IV (Caucasian) | Part 1: Sotrovimab 500 mg IV (Japanese) | Part 1: Sotrovimab 500 mg IV (Caucasian)
Number analyzed (Participants) | 3 | 3 | 9 | 9
Participants
  AST, High, Grade 0 to Grade 2 | 0 | 0 | 0 | 1
  Total Bilirubin, High, Grade 0 to Grade 1 | 1 | 1 | 0 | 0
  Total Bilirubin, High, Grade 0 to Grade 2 | 0 | 0 | 1 | 0
  Direct Bilirubin, High, Grade 0 to Grade 3 | 0 | 0 | 1 | 0
  Glucose (fasting), High, Grade 0 to Grade 1 | 0 | 0 | 0 | 3
  Glucose (fasting), High, Grade 0 to Grade 2 | 0 | 0 | 0 | 1
  Glucose, Low, Grade 1 to Grade 0 | 0 | 1 | 0 | 0
  Sodium, Low, Grade 0 to Grade 1 | 0 | 0 | 0 | 1

38. Secondary Outcome: Part 1: Number of Participants With Any Increase in Worst-case Urinalysis Results Post-Baseline Relative to Baseline by Dipstick Method Through Week 18
Description: Urine samples were collected for analysis of bilirubin, leukocyte esterase, occult blood and protein by a dipstick method. The dipstick test gives results in a semi-quantitative manner indicating proportional concentrations in the urine sample. Baseline is defined as the latest pre-dose assessment with a non-missing value on or after Day -1 visit, including those from unscheduled visits. Any increase means any increase to small, moderate, severe, potentially life threatening or positive post-Baseline relative to Baseline. Data is presented for only those parameters for which participants had any increase in urinalysis results post-Baseline relative to Baseline. Number of participants with worst case any increase in urinalysis results post-Baseline relative to Baseline has been presented.
Time Frame: Baseline (Day 1) and up to Week 18
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Placebo IV (Japanese) | Part 1:Placebo IV (Caucasian) | Part 1: Sotrovimab 500 mg IV (Japanese) | Part 1: Sotrovimab 500 mg IV (Caucasian)
Number analyzed (Participants) | 3 | 3 | 9 | 9
Participants
  Bilirubin | 1 | 0 | 2 | 0
  Leukocyte Esterase | 1 | 1 | 3 | 1
  Occult Blood | 1 | 0 | 4 | 3
  Protein | 1 | 0 | 1 | 1

39. Secondary Outcome: Part 2: Number of Participants With SAE and Common Non-SAE Through Week 18
Description: as for outcome 15
Time Frame: Up to Week 18
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Placebo IM (Japanese) | Part 2: Placebo IM (Caucasian) | Part 2: Sotrovimab 500 mg IM (Japanese) | Part 2: Sotrovimab 500 mg IM (Caucasian)
Number analyzed (Participants) | 2 | 2 | 10 | 10
Participants
  SAE | 0 | 0 | 0 | 0
  Non-SAE | 0 | 1 | 4 | 3

40. Secondary Outcome: Part 2: Number of Participants With AESI Through Week 18
Description: Adverse events of special interest (AESI) are relevant known toxicities of other therapeutic mAbs or signals observed in nonclinical programs of sotrovimab. AESI were defined as Injection-related reactions including hypersensitivity reactions, Hypersensitivity (SMQ narrow), Injection site reactions, Immunogenicity related adverse drug reactions (ADR) and AE potentially related to antibody-dependent enhancement of disease (ADE).
Time Frame: Up to Week 18
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Placebo IM (Japanese) | Part 2: Placebo IM (Caucasian) | Part 2: Sotrovimab 500 mg IM (Japanese) | Part 2: Sotrovimab 500 mg IM (Caucasian)
Number analyzed (Participants) | 2 | 2 | 10 | 10
Participants
  Injection related reaction including hypersensitivity | 0 | 0 | 0 | 0
  Hypersensitivity (SMQ narrow) | 0 | 0 | 0 | 0
  Injection Site Reaction | 0 | 0 | 1 | 0
  Immunogenicity related ADR | 0 | 0 | 0 | 0
  AE potentially related to ADE | 0 | 0 | 0 | 0

41. Secondary Outcome: Part 2: Number of Participants With Abnormal Clinically Significant ECG Findings Through Week 18
Description: Twelve 12-lead ECG's were obtained in the semi-recumbent or supine position after 10 minutes of rest using an ECG machine. Clinically significant abnormal findings are those which are not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition. Data for the number of participants with abnormal clinically significant worst case post-Baseline ECG findings were reported.
Time Frame: Up to Week 18
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Placebo IM (Japanese) | Part 2: Placebo IM (Caucasian) | Part 2: Sotrovimab 500 mg IM (Japanese) | Part 2: Sotrovimab 500 mg IM (Caucasian)
Number analyzed (Participants) | 2 | 2 | 10 | 10
Participants | 0 | 0 | 0 | 0

42. Secondary Outcome: Part 2: Number of Participants With Vital Signs Grade Shifts From Baseline Grade Through Week 18
Description: as for outcome 36
Time Frame: Baseline (Day 1) and up to Week 18
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Placebo IM (Japanese) | Part 2: Placebo IM (Caucasian) | Part 2: Sotrovimab 500 mg IM (Japanese) | Part 2: Sotrovimab 500 mg IM (Caucasian)
Number analyzed (Participants) | 2 | 2 | 10 | 10
Participants
  DBP; Grade 0 to Grade 1 | 0 | 0 | 1 | 0
  SBP; Grade 1 to Grade 0 | 0 | 0 | 1 | 0

43. Secondary Outcome: Part 2: Number of Participants With Clinical Chemistry Grade Shifts From Baseline Grade Through Week 18
Description: Blood samples were collected for analysis of clinical chemistry parameters including Alanine aminotransferase, Alkaline Phosphatase, Aspartate Aminotransferase, Total Bilirubin, Creatinine, Glucose (fasting), Glucose, Potassium and Sodium. Baseline is latest pre-dose assessment with a non-missing value on or after Day -1 visit including those from unscheduled visits. Grade Shift from Baseline is defined as shift from any grade (at Baseline) to Grades 1, 2, 3 and 4 post-Baseline. A worst post-Baseline grade shift is defined as worst change that occurred at any measured time point during treatment period. Grading was determined by the Division of Acquired Immunodeficiency Syndrome Table for Grading Severity (DAIDS) version 2.1. Grade 0=Normal, Grade 1=Mild, Grade 2=Moderate, Grade 3=Severe and Grade 4= Potentially Life-Threatening. Data is presented for only those parameters for which participants had grade shifts from Baseline grade. Worst-case post-Baseline shift data is presented.
Time Frame: Baseline (Day 1) and up to Week 18
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Placebo IM (Japanese) | Part 2: Placebo IM (Caucasian) | Part 2: Sotrovimab 500 mg IM (Japanese) | Part 2: Sotrovimab 500 mg IM (Caucasian)
Number analyzed (Participants) | 2 | 2 | 10 | 10
Participants
  ALT, High, Grade 0 to Grade 1 | 0 | 0 | 0 | 1
  ALP, High, Grade 0 to Grade 1 | 0 | 0 | 0 | 1
  AST, High, Grade 0 to Grade 1 | 0 | 0 | 1 | 0
  Total Bilirubin, High, Grade 0 to Grade 1 | 0 | 0 | 1 | 0
  Creatinine, High, Grade 0 to Grade 2 | 1 | 0 | 0 | 0
  Glucose (fasting), High, Grade 0 to Grade 2 | 0 | 0 | 1 | 0
  Glucose, Low, Grade 0 to Grade 1 | 1 | 0 | 0 | 1
  Potassium, High, Grade 0 to Grade 1 | 0 | 0 | 0 | 1
  Sodium, Low, Grade 0 to Grade 1 | 0 | 0 | 1 | 0
  Sodium, Low, Grade 1 to Grade 1 | 0 | 0 | 1 | 1

44. Secondary Outcome: Part 2: Number of Participants With Any Increase in Worst-case Urinalysis Results Post-Baseline Relative to Baseline by Dipstick Method Through Week 18
Description: Urine samples were collected for analysis of bilirubin, glucose, leukocyte esterase, nitrite, occult blood, protein and urobilinogen by a dipstick method. The dipstick test gives results in a semi-quantitative manner indicating proportional concentrations in the urine sample. Baseline is defined as the latest pre-dose assessment with a non-missing value on or after Day -1 visit, including those from unscheduled visits. Any increase means any increase to small, moderate, severe, potentially life threatening or positive post-Baseline relative to Baseline. Data is presented for only those parameters for which participants had any increase in urinalysis results post-Baseline relative to Baseline. Number of participants with worst case any increase in urinalysis results post-Baseline relative to Baseline has been presented.
Time Frame: Baseline (Day 1) and up to Week 18
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Placebo IM (Japanese) | Part 2: Placebo IM (Caucasian) | Part 2: Sotrovimab 500 mg IM (Japanese) | Part 2: Sotrovimab 500 mg IM (Caucasian)
Number analyzed (Participants) | 2 | 2 | 10 | 10
Participants
  Bilirubin | 1 | 0 | 1 | 0
  Glucose | 0 | 0 | 2 | 0
  Leukocyte Esterase | 0 | 1 | 3 | 2
  Nitrite | 0 | 0 | 1 | 0
  Occult Blood | 1 | 1 | 2 | 4
  Protein | 0 | 0 | 2 | 3
  Urobilinogen | 0 | 0 | 0 | 1

45. Other Pre Specified Outcome: Part 1 and Part 2: Bioavailability of Sotrovimab IM Versus IV Formulation Using AUClast
Description: Bioavailability of Sotrovimab was estimated using ANCOVA model with AUClast as dependent variable and ethnicity, body weight, route of administration as covariates with all available data (Part 1 [IV] and Part 2 [IM]) of Sotrovimab concentrations in serum. The AUClast Geometric Least Squares (LS) Means were estimated for each formulation and then a single parameter reported as the ratio of the AUClast geometric LS means (IM/IV) along with the 90% Confidence Interval were calculated. A single ratio parameter derived using the Geometric LS Means of AUClast IM versus IV and associated 90% Confidence Interval are presented.
Time Frame: Part 1: Day 1 (Pre-dose, at end of infusion and 1,2,6,8,24 [Day 2] and 48 [Day 3] hours after end of infusion); Weeks 2,3,4,6,8,12,18; Part 2: Day 1(Pre-dose and 1,2,6,8,24 [Day 2] and 48 [Day 3] hours after first IM injection); Weeks 2,3,4, 6,8,12,18
Population: Pharmacokinetic Population. Given that bioavailability assessment requires comparison of exposures between IM and IV routes of administration, data from Part 1 (IV) and Part 2 (IM) were combined to enable an estimation of bioavailability of IM formulation.
Measure: Number (90% Confidence Interval); unit: Ratio
Groups:
- Part 1 and Part 2: All Participants: In Part 1, Caucasian and Japanese participants were administered a single IV infusion of Sotrovimab at a dose of 500 mg on Day 1. In Part 2, Caucasian and Japanese participants were administered a single IM injection of Sotrovimab at a dose of 500 mg on Day 1.
Arm/Group | Part 1 and Part 2: All Participants
Number analyzed (Participants) | 38
Ratio | 0.5179 [0.4498 to 0.5964]

ADVERSE EVENTS:
Time Frame: All-cause mortality, serious adverse events (SAE) and non-serious adverse events (non-SAE) were collected up to Week 18 in Parts 1 and 2 of the study
Description: Safety Population was used to assess all-cause mortality, SAE and non-SAE which comprised of all randomized participants who were exposed to study intervention.
Arm/Group | Part 1: Placebo IV (Japanese) | Part 1:Placebo IV (Caucasian) | Part 1: Sotrovimab 500 mg IV (Japanese) | Part 1: Sotrovimab 500 mg IV (Caucasian) | Part 2: Placebo IM (Japanese) | Part 2: Placebo IM (Caucasian) | Part 2: Sotrovimab 500 mg IM (Japanese) | Part 2: Sotrovimab 500 mg IM (Caucasian)
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/9 | 0/9 | 0/2 | 0/2 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/9 | 0/9 | 0/2 | 0/2 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 1/3 | 1/3 | 2/9 | 1/9 | 0/2 | 1/2 | 4/10 | 3/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Placebo IV (Japanese) (N=3) | Part 1:Placebo IV (Caucasian) (N=3) | Part 1: Sotrovimab 500 mg IV (Japanese) (N=9) | Part 1: Sotrovimab 500 mg IV (Caucasian) (N=9) | Part 2: Placebo IM (Japanese) (N=2) | Part 2: Placebo IM (Caucasian) (N=2) | Part 2: Sotrovimab 500 mg IM (Japanese) (N=10) | Part 2: Sotrovimab 500 mg IM (Caucasian) (N=10)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — General disorders and administration site conditions
Feeling hot (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) — General disorders and administration site conditions
Injection site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — General disorders and administration site conditions
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Sleep paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nightmare (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vascular pain (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-05-27): https://cdn.clinicaltrials.gov/large-docs/52/NCT04988152/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-09): https://cdn.clinicaltrials.gov/large-docs/52/NCT04988152/SAP_001.pdf